CLINICAL TRIAL: NCT04066140
Title: Patient Activation in Incident Dialysis
Brief Title: Patient Activation in Dialysis
Acronym: PAMD
Status: Completed | Type: Observational
Sponsor: Satellite Healthcare (Other)
Responsible Party: Sponsor
Other Study IDs: SIH118PAMD
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2019-08

CONDITIONS: Renal Dialysis; Kidney Failure, Chronic
Keywords: patient activation; self management
MeSH Terms: conditions — Kidney Failure, Chronic; Patient Participation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No Intervention. Observational Study.

SUMMARY:
Patient activation refers to patients' willingness and ability to make independent actions to manage their health and care and requires knowledge, skill and confidence. This study aims to explore activation levels of incident dialysis patients at start of dialysis and after 3 months of dialysis.

DETAILED DESCRIPTION:
Patient activation refers to patients' willingness and ability to make independent actions to manage their health and care and requires knowledge, skill and confidence. This study aims to explore activation levels, using the 13 item PAM-13 survey, of incident dialysis patients at start of dialysis and after 3 months of dialysis.

ELIGIBILITY:
Inclusion Criteria:

-Incident dialysis patients commencing at Satellite Healthcare during study recruitment dates

Exclusion Criteria:

* Age < 18 years
* Started dialysis more than 3 weeks prior to identification
* Transitioning to dialysis at a participating center from a non-participating center, when that patient has been on dialysis for more than 3 weeks at any center.
* Transitioning to dialysis after kidney transplant failure
* Inability to participate because of cognitive impairment or active psychological condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Incident dialysis patients commencing at Satellite Healthcare
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2019-12-08 (Actual); Study Completion 2020-06-17 (Actual)

PRIMARY OUTCOMES:
Patient Activation | 3 months
  Patient Activation as measured by PAM-13 instrument

CONTACTS AND LOCATIONS:
Overall Officials: Wael Hussein, MD, Principal Investigator — Satellite Healthcare
Locations (36):
- United States (36):
  - Satellite Dialysis Daly City, Daly City, California
  - Satellite Healthcare Los Gatos, Los Gatos, California
  - Satellite Healthcare Merced, Merced, California
  - Satellite Healthcare Central Modesto, Modesto, California
  - WellBound Modesto, Modesto, California
  - Satellite Healthcare Modesto, Modesto, California
  - WellBound North Modesto, Modesto, California
  - Satellite Dialysis Morgan Hill, Morgan Hill, California
  - Satellite Healthcare Oakland, Oakland, California
  - Satellite Healthcare Orange, Orange, California
  - Satellite Healthcare Rohnert Park, Rohnert Park, California
  - Satellite Wellbound Sacramento, Sacramento, California
  - Satellite Healthcare Sacramento, Sacramento, California
  - Satellite Healthcare San Carlos, San Carlos, California
  - Satellite Healthcare San Francisco, San Francisco, California
  - WellBound San Francisco, San Francisco, California
  - Satellite Dialysis Silver Creek, San Jose, California
  - Wellbound San Jose, San Jose, California
  - Satellite Healthcare, San Jose, California
  - Satellite Dialysis West San Leandro, San Leandro, California
  - Satellite Healthcare Santa Ana, Santa Ana, California
  - WellBound Santa Rosa, Santa Rosa, California
  - WellBound Stockton, Stockton, California
  - Satellite Dialysis Sunnyvale, Sunnyvale, California
  - Satellite Healthcare Tracy, Tracy, California
  - Satellite Healthcare Turlock, Turlock, California
  - WellBound Vallejo, Vallejo, California
  - Satellite Dialysis Watsonville, Watsonville, California
  - Satellite Healthcare Poplar, Memphis, Tennessee
  - Satellite Healthcare Chickasaw Gardens, Memphis, Tennessee
  - WellBound Memphis, Memphis, Tennessee
  - Satellite Healthcare Metric, Austin, Texas
  - Wellbound Austin, Austin, Texas
  - Satellite Healthcare Kyle, Kyle, Texas
  - Satellite Healthcare Laredo South, Laredo, Texas
  - Satellite Healthcare Round Rock, Round Rock, Texas

IPD SHARING:
Plan to Share IPD: No
Overall findings will be disseminated through publications and conference presentations.